CLINICAL TRIAL: NCT02407119
Title: Effect of Helicobacter Pylori Eradication on Glandular Atrophy and Metachronous Cancer in Patients Undergoing Endoscopic Mucosal Resection for Gastric Cancer
Brief Title: Effects of H. Pylori Eradication on the Gastric Preneoplastic Lesion and Neoplasm After ESD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Il Ju Choi, MD, PhD, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCCCTS03-062; 1310280 (Other Grant/Funding Number: National Cancer Center, Korea)
Record Dates: First submitted 2015-03-13; First posted 2015-04-02 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Helicobacter Pylori Infection; Early Gastric Cancer; Endoscopic Resection
Keywords: H. pylori eradication; Atrophy; Intestinal metaplasia; Endoscopic resection; Stomach neoplasm
MeSH Terms: conditions — Stomach Neoplasms; Atrophy | interventions — Rabeprazole; Clarithromycin; Amoxicillin; Proton Pump Inhibitors; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 7 day H.pylori eradication (Active Comparator): Treatment: Omeprazole 20 mg or Rabeprazole 10 mg bid + clarithromycin 500 mg and amoxicillin 1,000 mg bid for 7 days
  Interventions: Drug: 7 day H.pylori eradication Omeprazole or Rabeprazole, Clarithromycin, Amoxicillin
- Placebo (Placebo Comparator): Omeprazole 20 mg or Rabeprazole 10 mg bid + Placebo for two antibiotics (clarithromycin and amoxicillin) bid for 7 days
  Interventions: Drug: Placebo, Omeprazole or Rabeprazole, Clarithromycin

INTERVENTIONS:
Drug: 7 day H.pylori eradication Omeprazole or Rabeprazole, Clarithromycin, Amoxicillin — Omeprazole 20 mg or Rabeprazole 10 mg bid for 7 days, Clarithromycin 500 mg bid for 7 days, Amoxicillin 1,000 mg bid for 7 days.
  Other Names: 7 day Proton pump inhibitor (PPI)-based standard triple therapy
  Arms: 7 day H.pylori eradication
Drug: Placebo, Omeprazole or Rabeprazole, Clarithromycin — Omeprazole 20 mg or Rabeprazole 10 mg bid for 7 days, Placebo for clarithromycin 500 mg bid for 7 days, Placebo for amoxicillin 1,000 mg bid for 7 days.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates whether Helicobacter pylori eradication improves precancerous lesions including glandular atrophy and intestinal metaplasia as well as metachronous cancers or dysplasias after endoscopic mucosal resection for gastric cancer.

DETAILED DESCRIPTION:
Helicobacter pylori is a primary etiological agent leading to chronic gastritis and peptic ulcer. The organism is also associated with gastric cancer in epidemiological studies. However detailed mechanism of carcinogenesis remains unknown. Histolopathological studies indicate that chronic H. pylori infection progresses over decades through stages of chronic gastritis, atrophy, intestinal metaplasia, dysplasia and cancer. Gastric atrophy and intestinal metaplasia are considered as precancerous lesions, but whether H. pylori eradication improves these lesions and prevents metachronous gastric cancer is controversial. And the issue has not been evaluated in gastric cancer patients. However, despite the conflicting evidences from two open labelled randomized controlled trials, current guidelines from various regions recommend H. pylori eradication treatment in patients who were treated for gastric cancer by surgically or endoscopically. Thus, it is important to evaluate whether H. pylori eradication can improve known precancerous lesion, i.e. glandular atrophy and intestinal metaplasia in gastric cancer patients. Such histological improvement can eventually reduce secondary gastric cancer development and provide evidence for current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Early Gastric cancer or high grade dysplasia confirmed by endoscopy

  * Histologically confirmed well or moderately differentiated adenocarcinoma, or high grade dysplasia
  * Submucosal invasion is not suspected
  * No evidence of ulceration or ulcer scar within the lesion
* Helicobacter pylori infection was confirmed by histological evaluation and rapid urease test
* Pre op CT stage: IA (T1N0M0) according to UICC TNM classification system
* Informed consent should be signed

Exclusion Criteria:

* Recurrent gastric cancer
* Previous serious side effect to antibiotics
* H. pylori eradication treatment history
* Poorly differentiated adenocarcinoma or Signet ring cell carcinoma
* Undergoing operation due to complication of EMR
* Undergoing operation due to remnant cancer
* Other malignancy within the past 5 years
* Pregnant or nursing women
* Serious concurrent infection or nonmalignant disease such as liver cirrhosis, renal failure, cardiovascular diseases
* Psychiatric disorder that would preclude compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Improvement (histological) of glandular atrophy | 3 years after enrollment
  Improvement of glandular atrophy at the corpus lesser curvature
Incidence of metachronous gastric cancer | 3 years after last patient enrollment
  Comparison of metachronous gastric cancer according to the allocated treatment

SECONDARY OUTCOMES:
Incidence of new gastric dysplasia | 3 years after last patient enrollment
  Comparison of new gastric dysplasia according to the allocated treatment
Overall survival | 3 years after last patient enrollment
  Comparison of overall survival according to the allocated treatment

CONTACTS AND LOCATIONS:
Overall Officials: Il Ju Choi, MD, PhD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi IJ, Kook MC, Kim YI, Cho SJ, Lee JY, Kim CG, Park B, Nam BH. Helicobacter pylori Therapy for the Prevention of Metachronous Gastric Cancer. N Engl J Med. 2018 Mar 22;378(12):1085-1095. doi: 10.1056/NEJMoa1708423. PMID 29562147